CLINICAL TRIAL: NCT01958086
Title: Visuomotor Prosthetic for Paralysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Richard A. Andersen, PhD (Other)
Collaborators: University of California, Los Angeles (Other); Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Sponsor-Investigator, Richard A. Andersen, PhD, James G. Boswell Professor of Neuroscience, California Institute of Technology
Organization: California Institute of Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: G120287; 13-000576 (Other: UCLA IRB application number)
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Quadriplegia
Keywords: Neural; Prosthetic; brain machine interface; brain computer interface; brain control; paralysis; tetraplegia; quadriplegia; spinal cord injury
MeSH Terms: conditions — Quadriplegia; Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neural Communication System (Experimental): The Neural Communication System consists of two Neuroport Multi-Port Arrays, which are descried in detail in the intervention description. One Neuroport Multi-Port Array is inserted into the posterior parietal cortex, an area of the brain used in reach planning. The second Neuroport Multi-Port Array is inserted into the motor cortex, which is primarily responsible for controlling movement. The arrays are inserted and the percutaneous pedestal is attached to the skull during a surgical procedure. Following surgical recovery the subject will participate in study sessions 3-5 times per week in which they will learn to use thought to control a simple computer environment or a tablet computer.
  Interventions: Device: Neural Communication System

INTERVENTIONS:
Device: Neural Communication System — NeuroPort Arrays allow for the local recording of cerebral cortex. The Neural Communication system is primarily composed of two NeuroPort Arrays. The two arrays of one MultiPort device will be placed in the primary motor cortex for recording (Platinum-tipped electrodes); and the two arrays of the additional MultiPort device be placed in the superior parietal lobule for recording (Platinum-tipped electrodes). Each MultiPort device consists of two arrays, each with 100 electrodes in a 10 x 10 configuration, with dimensions 4 mm x 4 mm x 1.5 mm (W x H x D) or 4 mm x 4 mm x 1.0 mm, and a titanium percutaneous connector, 19 mm diameter at the base. Each MultiPort can have a total of 128 active channels (capable of transmitting neural signals to the percutaneous connector) across the two arrays. In our design, we will split active channels evenly between the two arrays resulting in 64 active channels per array.
  Other Names: NeuroPort Multi-Port Array

SUMMARY:
The investigators objective is to run human clinical trials in which brain activity recorded through a "brain-chip" implanted in the human brain can be used to provide novel communication capabilities to severely paralyzed individuals by allowing direct brain-control of a computer interface. A prospective, longitudinal, single-arm early feasibility study will be used to examine the safety and effectiveness of using a neural communication system to control a simple computer interface and a tablet computer. Initial brain control training will occur in simplified computer environments, however, the ultimate objective of the clinical trial is to allow the human patient autonomous control over the Google Android tablet operating system. Tablet computers offer a balance of ease of use and functionality that should facilitate fusion with the BMI. The tablet interface could potentially allow the patient population to make a phone call, manage personal finances, watch movies, paint pictures, play videogames, program applications, and interact with a variety of "smart" devices such as televisions, kitchen appliances, and perhaps in time, devices such as robotic limbs and smart cars. Brain control of tablet computers has the potential to greatly improve the quality of life of severely paralyzed individuals. Five subjects will be enrolled, each implanted with the NCS for a period of at least 53 weeks and up to 313 weeks. The study is expected to take at least one year and up to six years in total.

DETAILED DESCRIPTION:
The objective of the proposed research is to obtain scientific knowledge of visuomotor transformations in posterior parietal cortex (PPC) and primary motor cortex (M1) from tetraplegic subjects in a clinical trial to advance the development of neural prosthetics. We have shown in clinical trials conducted over the past 6 years that PPC can control neural prosthetics for assisting tetraplegic subjects. Other groups have concentrated on M1 and likewise find control for neural prosthetics. In our studies of PPC we have found that besides trajectory signals to move robotic limbs or control computer cursors, there are a plethora of visuomotor signals that represent intended movements of most of the body, movement goals, cognitive strategies, and even memory signals. Our central hypothesis is that PPC and M1 will encode visuomotor parameters in both similar and different ways, and that algorithms can be developed to leverage those signals from the two areas that are complimentary to improve prosthetic range and performance. Implants will be made in both M1 and PPC, enabling simultaneous recording in the same subjects, elevating concerns of comparing data from different labs collected in different individuals with different implants and different tasks.

This central hypothesis will be tested in two broad aims, for which we have substantial preliminary data. Aim 1 will examine the control of the body by the two areas. It is hypothesized that M1 will demonstrate strong specificity for the contralateral limb (implants will be made in the hand knob) whereas PPC will code movements for most of the body and on both contra and ipsilateral sides by leveraging its partially mixed encoding of parameters (subaim 1a). Whereas M1 is hypothesized to code spatial variables exclusively during attempted or imagined actions, it is hypothesized that PPC also encodes cognitive spatial variables in task appropriate reference frames (subaim 1b). In subaim 1c we will examine how multiple body parts are combined in movement representations, hypothesizing that M1 and PPC will employ a diverse set of mechanisms including linear summation, non-linear combinations, and movement suppression expressed in different ways as a function of brain area and the specific movement set.

Aim 2 will examine the temporal aspects of encoding in the two areas. In subaim 2a we will test the hypothesis that the neural dynamics during sustained periods of movement are largely unchanging in both areas. In subaim 2b we hypothesize that, during sequential movements, M1 codes only the ongoing movement whereas PPC codes both the current and subsequent movements. Finally, in subaim 2c we will examine the coding of movement speed, with the hypothesis that there are separate subspaces in both M1 and PPC for direction and speed of movement.

ELIGIBILITY:
Inclusion Criteria:

* Pathology resulting in paralysis
* Age 22-65 years
* Able to provide informed consent
* Understand and comply with instructions, if necessary, with the aid of a translator
* Able to communicate via speech
* Surgical clearance
* Life expectancy greater than 12 months
* Live within 60 miles of study location and willing to travel up to 5 days per week
* A regular caregiver to monitor the surgical site
* Psychosocial support system
* Stable ventilator status

Exclusion Criteria:

* Intellectual impairment
* Psychotic illness or chronic psychiatric disorder, including major depression if untreated
* Poor visual acuity
* Pregnancy
* Active infection or unexplained fever
* Scalp lesions or skin breakdown
* HIV or AIDS infection
* Active cancer or chemotherapy
* Medically uncontrolled diabetes
* Autonomic dysreflexia
* History of seizure
* Implanted hydrocephalus shunt
* History of supratentorial brain injury or neurosurgery
* Medical conditions contraindicating surgery and chronic implantation of a medical device
* Unable to undergo MRI or anticipated need for MRI during study
* Nursing an infant or unwilling to bottle-feed infant
* Chronic oral or intravenous use of steroids or immunosuppressive therapy
* Suicidal ideation
* Drug or alcohol dependence
* Planning to become pregnant, or unwilling to use adequate birth control
* Implanted Cardiac Defibrillator, Pacemaker, vagal nerve stimulator, or spinal cord stimulator.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Subject control of a tablet computer | Six years after array implantation
  Assessments will be compared with chance and previous reports of BMI efficacy using control signals derived from primary motor cortex. Computer-interface competency examination that measures the ability of the subject to control various aspects of the tablet user interface. Additionally we will measure the Quality of Life Inventory (QOLI) at regular intervals over the duration of the study. Changes in performance over time.
Absence of infection or irritation | Six years after array implantation
  The Serious Adverse event (SAE) rate will be calculated as the number of SAEs per implant-days. The SAE rate will be continuously compared to the 1% threshold level. CT scan; inspection of patient's scalp for evidence of reddening or discharge; review of new symptoms including possible fever, headache, visual or auditory changes, or change in mood or behavior; serial neurologic exams. The condition of the area will be compared with its condition on previous visits. History will be obtained regarding new symptoms.
  Neurologic exam will be compared to baseline neurologic exam

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Andersen, PhD, Principal Investigator — California Institute of Technology; Ausaf Bari, MD, PhD, Principal Investigator — University of California, Los Angeles; Emily Rosario, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (3):
- United States (3):
  - University of California Los Angeles, Los Angeles, California
  - California Institute of Technology, Pasadena, California
  - Casa Colina Centers for Rehabilitation, Pomona, California

REFERENCES:
- [Derived] Bashford L, Rosenthal IA, Kellis S, Bjanes D, Pejsa K, Brunton BW, Andersen RA. Neural subspaces of imagined movements in parietal cortex remain stable over several years in humans. J Neural Eng. 2024 Aug 28;21(4):046059. doi: 10.1088/1741-2552/ad6e19. PMID 39134021
- [Derived] Guan C, Aflalo T, Zhang CY, Amoruso E, Rosario ER, Pouratian N, Andersen RA. Stability of motor representations after paralysis. Elife. 2022 Sep 20;11:e74478. doi: 10.7554/eLife.74478. PMID 36125116